CLINICAL TRIAL: NCT02283450
Title: Regulation of Immunological Cytokines by Qiliqiangxin Capsule in Dilated Cardiomyopathy patients--a Randomized Double Blind Clinical Trial
Brief Title: Regulation of Immunological Cytokines by Qiliqiangxin Capsule in Dilated Cardiomyopathy Patients
Status: Completed | Type: Observational
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Wei Liu, Prof., Harbin Medical University
Other Study IDs: 2013
Record Dates: First submitted 2014-11-02; First posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — qiliqiangxin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- the experimental group: The patients in experimental group received the relevant tests and inspections before the beginning of experiment，signed the informed consent. Then we get the venous blood centrifugalization and cryopreservation. The patients take the medicine qiliqiangxin three times per day，four tablets at a time. Afrer a month，we evaluated the symptoms，the function of heart，blood pressure，heart rate and keep blood specimens. Three and six month later，electrocardiogram and echocardiography were taken and the determination of the NT - proBNP was done.
  Interventions: Drug: Qiliqiangxin Capsule
- the placebo group: The placebo group was followed up in the same way.
  Interventions: Drug: Qiliqiangxin Capsule

INTERVENTIONS:
Drug: Qiliqiangxin Capsule

SUMMARY:
Purpose :Research into the impact of Qiliqiangxin capsule on IFN-γ，IL-4，NT-proBNP in dilated cardiomyopathy patients with heart failure.

Methods :Data were collected from the patients with idiopathic dilated cardiomyopathy ( cardiac function NYHA Ⅱ-Ⅳ) in the first affiliated hospital of Harbin Medical University from May 2012 to April 2014. These 30 cases were treated under the recommendations of normal diagnosis and treatment in cardiomyopathy. This experiment was randomized double-blinded，the experimental interferences were avoided and patients were divided into the experimental group and the placebo group. The patients in experimental group received the relevant tests and inspections before the beginning of experiment，signed the informed consent. Then the investigators get the venous blood centrifugalization and cryopreservation. The patients take the medicine qiliqiangxin three times per day，four tablets at a time. Afrer a month，the investigators evaluated the symptoms，the function of heart，blood pressure，heart rate and keep blood specimens. Three and six month later，electrocardiogram and echocardiography were taken and the determination of the NT - proBNP was done. The placebo group was followed up in the same way.

ELIGIBILITY:
Inclusion Criteria:

* Congetive heart failure

Exclusion Criteria:

* Valvular heart diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: congestive heart failure.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
cytokine level at 3 months | 3 months